CLINICAL TRIAL: NCT01756612
Title: A Non-interventional Study to Assess the Hemoglobin Level Depending on the Comorbidity Index in Chronic Kidney Disease (CKD) Patients Not in Dialysis Treated With Mircera®
Brief Title: A Study to Assess Hemoglobin Level Depending on the Comorbidity Index in Chronic Kidney Disease (CKD) Participants Not in Dialysis Treated With Methoxy Polyethylene Glycol-Epoetin Beta (COMETE)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28145
Record Dates: First submitted 2012-12-19; First posted 2012-12-27 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Renal Anemia of Chronic Kidney Disease
MeSH Terms: interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Chronic Kidney Disease Participants: Participants for whom the treating physician has decided to initiate treatment with MIRCERA for medical reasons prior to study start, will be observed for 9 months.
  Interventions: Drug: Methoxy Polyethylene Glycol-Epoetin Beta

INTERVENTIONS:
Drug: Methoxy Polyethylene Glycol-Epoetin Beta — Methoxy polyethylene glycol-epoetin beta will be administered at the discretion of treating physician. Study protocol does not specify any treatment regimen.
  Other Names: Mircera

SUMMARY:
This prospective, multicenter, observational study will evaluate the impact of comorbidity factors on the hemoglobin level in participants with chronic kidney disease who are not on dialysis and initiated on treatment with methoxy polyethylene glycol-epoetin beta (Mircera). Data will be collected for 9 months after initiation of methoxy polyethylene glycol-epoetin beta treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic kidney disease not on dialysis
* Treatment-naïve for erythropoiesis-stimulating agents (ESAs), not having received ESAs in the 6 months prior to inclusion in this study
* Hemoglobin level less then (<)10 grams per deciliter (g/dL) at inclusion
* Participants for whom the treating physician has decided to initiate treatment with methoxy polyethylene glycol-epoetin beta for medical reasons prior to study start

Exclusion Criteria:

* Functional renal transplant
* Current participation in a clinical trial in anemia due to chronic kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ESA naïve participants with chronic kidney disease who are not on dialysis
Sampling Method: Non-Probability Sample
Enrollment: 551 (Actual)
Dates: Start 2012-11-21 (Actual); Primary Completion 2015-03-25 (Actual); Study Completion 2015-03-25 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With an Increase From Baseline in Hemoglobin Level of Greater Than or Equal to (>/=) 1 g/dL or a Hemoglobin Level Between 10 and 12 g/dL After 9 Months of Treatment Without any Transfusional Recourse | Baseline, Month 9

SECONDARY OUTCOMES:
Hemoglobin Levels According to Liu Index and Resistance Factors | Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9
Average Dose of Mircera in Total Population | Baseline up to 9 months
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) in Total Population | Baseline up to 9 months
Average Dose of Mircera in Subgroups as Defined by the Comorbidities List Used for the Charlson Comorbidities Index Calculation | Baseline up to 9 months
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) in in Subgroups as Defined by the Comorbidities List Used for the Charlson Comorbidities Index Calculation | Baseline up to 9 months
Duration of Treatment With Mircera | Baseline up to 9 months
Number of Participants Who Received Concomitant Treatment (Known as Potentially Resistant Factors) for Renal Anemia | Baseline up to 9 month

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (108):
- France (108):
  - CHP Aix, Aix-en-Provence
  - Ch Notre Dame Misericorde; Hemodialyse, Ajaccio
  - Chi D Alencon;Nephrologie Hemodialyse, Alençon
  - Centre Aider, Alès
  - Hotel Dieu; Nephrologie Hemodialyse, Angers
  - Centre Hospitalier; Hemodialyse, Annonay
  - Centre Hemodialyse La Riviera, Antibes
  - Ch D Arras; Nephrologie, Arras
  - Chp Aubagne, Aubagne
  - Ch Henri Duffaut; Nephrologie Hemodialyse, Avignon
  - Chic Cote Basque Bayonne; Nephrologie Hemodialyse, Bayonne
  - Ch De Beauvais; Neph Endocrino Dialyse Diabeto, Beauvais
  - Centre D Hemodialyse Regina, Belley
  - CHU Saint Jacques; Centre De Dialyse, Besançon
  - Ch Germon Et Gauthier; Medecine Interne Nephrologie, Beuvry
  - CNB - Centre Nephrologie Du Biterrois, Béziers
  - Centre Hemodialyse St Augustin; Nephrologie, Bordeaux
  - Hopital Pellegrin; Departement Nephrologie, Bordeaux
  - Cabinet Medical, Bordeaux
  - Ch De Fleyriat; Nephrologie Hemodialyse, Bourg-en-Bresse
  - Aural; Service Hemodialyse, Bourgoin
  - Hopital La Cavale Blanche; Nephrologie, Brest
  - Ch de Brive la Gaillarde; Nephrologie Hemodialyse, Brive-la-Gaillarde
  - Centre D Hemodialyse Saint Roch, Cabestany
  - Hopital Clemenceau; Nephrologie Hemodialyse, Caen
  - Ch Antoine Gayraud; Nephrologie Hemodialyse, Carcassonne
  - Centre Hemodialyse Du Lez; Nephrologie, Castelnau-le-Lez
  - CH William Morey; Nephrologie, Chalon-sur-Saône
  - Aura Auvergne; Aura Auvergne, Chamalières
  - Ch De Chambery; Nephrologie, Chambéry
  - Avitum France; Centre De Nephrologie, Châteauroux
  - Centre Hospitalier; Hemodialyse, Cholet
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - Centre De Sante Medical; Centre De Sante Republique, Clermont-Ferrand
  - Ch Laennec; Nephrologie Hemodialyse, Creil
  - Fondation Transplantation; Ctirc De Drevon, Dijon
  - Nephrocare Ile De France; Etampes, Étampes
  - Chi Eure Seine D Evreux; Nephrologie, Évreux
  - Cabinet Medical, Fontaine-lès-Dijon
  - Hopital De Freyming; Nephrologie, Freyming-Merlebach
  - Centre Hospitalier General; Service de Nephrologie-Hemodialyse, Gap
  - Association Aurad Aquitaine; Aurad Gradignan, Gradignan
  - Centre de Dialyse Atirra; Service Nephrologie - Hemodialyse, Greize
  - Ch Dptal Les Oudairies; Nephrologie, La Roche-sur-Yon
  - Hopital Albert Michallon; Clinique De Nephrologie, La Tronche
  - Agduc Muller, La Tronche
  - Ch De Laon; Nephrologie Hemodialyse, Laon
  - Hopital Prive De L Estuaire; Nephrologie Hemodialyse, Le Havre
  - Ch Emile Roux; Nephrologie, Le Puy-en-Velay
  - Hopital Claude Huriez; Nephrologie, Lille
  - Polyclinique De La Louviere; Nephrologie, Lille
  - Ctre Hosp St Joseph Et St Luc; Nephrologie Hemodialyse, Lyon
  - Hopital Edouard-Herriot; Nephrologie - Hemodialyse, Lyon
  - Clinique Bouchard ; Nephrologie, Marseille
  - Hopital De La Conception; Hemodialyse, Marseille
  - Hopital De La Conception; Nephrologie, Marseille
  - Ch De Meaux; Medecine C, Meaux
  - Hopital Layne; Nephrologie Hemodialyse, Mont-de-Marsan
  - Hopital Hotel Dieu; Medecine Geriatrique Nephrologie, Mont-Saint-Martin
  - Centre D Hemodialyse Sodetir, Montereau
  - Centre Aider; Centre Aider Montpellier, Montpellier
  - Centre De Dialyse La Fonderie, Mullhouse
  - Polyclinique De Gentilly; Hemodialyse, Nancy
  - Hopital Hotel Dieu Et HME; Nephrologie Immunologie Clinique, Nantes
  - Hopital Hotel Dieu Et Hme; Hemodialyse Chronique, Nantes
  - Echo Nantes Confluent; Uad Montfort, Nantes
  - Hopital Pasteur; Pavillon A Nephrologie, Nice
  - Centre Gardialyse, Nîmes
  - Ctre Dialyse De La Reine Blanche, Orléans
  - Hopital de La Source; Service de Nephrologie & Hemodialyse, Orléans
  - Hopital Saint Louis; Service de Nephrologie - Transplantation, Paris
  - Ch Pitie Salpetriere; Nephrologie Hemodialyse, Paris
  - Hopital Europeen Georges Pompidou; Service de Nephrologie, Paris
  - Hopital Tenon; Nephrologie Dialyse, Paris
  - Hopital Saint Jean; Nephrologie, Perpignan
  - Centre Hemodialyse Saint Martin, Pessac
  - Ch Lyon Sud; Nephrologie Sect Jules Courmont, Pierre-Bénite
  - Chi Poissy Saint Germain En Laye; Hemodialyse, Poissy
  - Chu La Miletrie;Nephrologie Transplantation, Poitiers
  - Association Pour L'Aide Des Uremiques de Bretagne, Quimper
  - Hopital Pontchaillou; Nephrologie, Rennes
  - Clinique De L Europe; Hemodialyse, Rouen
  - Chi Du Val D Ariege; Gastro Enterologie Nephrologie, Saint-Jean-de-Verges
  - Centre D Hemodialyse, Saint-Laurent-du-Var
  - Centre D'Hemodialyse Arnaud Tzanck; Service Nephrologie - Hemodialyse, Saint-Laurent-du-Var
  - Institut Arnault Tzanck; Med 2, Saint-Laurent-du-Var
  - Memorial France Etats Unis; Nephrologie, Saint-Lô
  - Artic; Bureau, Saint-Priest-en-Jarez
  - Hopital Nord; Hopital De Jour, Saint-Priest-en-Jarez
  - HOPITAL NORD; NEPH Transplantation Reanimation, Saint-Priest-en-Jarez
  - Nephrocare Tassin Charcot; Nephrologie, Sainte-Foy-lès-Lyon
  - Hopital Sud ; Nephrologie Hemodialyse, Salouël
  - Centre Hospitalier De Sens; Nephrologie-Dialyse, Sens
  - Ch Gaston Ramon; Nephrologie, Sens
  - Ch De Soissons; Medecine 5, Soissons
  - Hopital Broussais; Medecine 4, St-Malo
  - Hopital Civil; Nephrologie Clinique Medicale B, Strasbourg
  - Nephrocare Ile de France; Suresnes, Suresnes
  - Hopital Foch; Nephrologie Hemodialyse, Suresnes
  - Hopital de La Gespe; Dept of Nephrology, Tarbes
  - Hopitaux Du Leman Site Thonon;Nephrologie, Thonon-les-Bains
  - Hopital Sainte Musse; Nephrologie, Toulon
  - Hopital Rangueil; Nephrologie Hemodialyse, Toulouse
  - Clinique de Tournan; Service de Nephrologie, Tournan-en-Brie
  - Hopital Bretonneau; Nephrologie Transplantations, Tours
  - Ch Bretagne Atlantique De Vannes; Nephrologie, Vannes
  - Hopital Saint Nicolas; Medecine A, Verdun
  - Cabinet Medical, Villeurbanne